CLINICAL TRIAL: NCT01744197
Title: Effect of Synera in Reducing Pain Associated With Venipuncture and Superficial Dermatologic Procedures
Brief Title: Synera Venipuncture Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12112
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Pain; Phlebotomy; Palliative Care
Keywords: Pain control; Needle stick pain; Venipuncture pain
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): First application: Synera (lidocaine 70mg/tetracaine 70mg) patch; Second application: Placebo patch
  Interventions: Drug: Synera (lidocaine 70mg/tetracaine 70mg)
- Arm 2 (Experimental): First application: Placebo patch; Second application: Synera (lidocaine 70mg/tetracaine 70mg) patch
  Interventions: Drug: Synera (lidocaine 70mg/tetracaine 70mg)

INTERVENTIONS:
Drug: Synera (lidocaine 70mg/tetracaine 70mg) — All subjects will receive 2 patch applications during this study: one Synera, one placebo. The 2 patch applications must be done on separate days. Only 1 patch will be used per application. Arm 1 subjects will receive Synera patch for the 1st application, and placebo for the second. Arm 2 patients will receive placebo patch for the 1st application, and Synera patch for the second.
  Other Names: Synera

SUMMARY:
Synera, which is a heated topical patch containing both lidocaine and tetracaine, is intended to reduce the pain associated with venipuncture and superficial dermatologic procedures by numbing the skin. This study will test the effectiveness of the Synera lidocaine/tetracaine patch when administered for 30 ± 5 minutes to provide dermal anesthesia in adult oncology patients undergoing venipuncture as part of their care, for treatment or diagnostics (laboratory or imaging). Compared to the use of the placebo patch, this study hypothesizes that the difference of 1 cm on the 0-10 visual analogue scale (VAS) will be observed 30 minutes after the use of the Synera patch. Pain intensity will be assessed by a 0-10 VAS

ELIGIBILITY:
Inclusion Criteria:

* Patients with any tumor type where treatment is received through venipuncture or any procedure that is needle based or who require regular pharmacokinetic (PK) study.
* Is 18 years of age or older.
* Patients expected to undergo the first venipuncture procedure within 5 working days of enrollment.
* Male or female patients
* Has signed the most recent Patient Informed Consent Form
* Has signed a Patient Authorization Form (HIPPA)

Exclusion Criteria:

* Patients with sensitivity to lidocaine, tetracaine, or any other component of the product
* Known sensitivity to any components of test materials (sulphites and adhesives)
* Patients with damaged or broken skin at the designated patch site
* Pregnant or breastfeeding women patients
* Use of any immediate-release single-agent opioid product (ie, morphine, oxycodone, hydrocodone, hydromorphone, oxymorphone, or tramadol) or combination products containing acetaminophen or ibuprofen with one of these agents within 4 hours of the patient's visit
* Previous irradiation to the site of the patch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Matson, RN, BSN, Principal Investigator — US Oncology Research, McKesson Specialty Health; Laura T. Guerra, RN, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 19 Locations Including, Dallas, Texas, United States

REFERENCES:
- [Result] Wallace MS, Kopecky EA, Ma T, Brophy F, Campbell JC. Evaluation of the depth and duration of anesthesia from heated lidocaine/tetracaine (Synera) patches compared with placebo patches applied to healthy adult volunteers. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):507-13. doi: 10.1097/AAP.0b013e3181fa69b8. PMID 20975464
- [Result] Sawyer J, Febbraro S, Masud S, Ashburn MA, Campbell JC. Heated lidocaine/tetracaine patch (Synera, Rapydan) compared with lidocaine/prilocaine cream (EMLA) for topical anaesthesia before vascular access. Br J Anaesth. 2009 Feb;102(2):210-5. doi: 10.1093/bja/aen364. PMID 19151049

RESULTS

PARTICIPANT FLOW:
Groups:
- Synera First, Then Placebo: Synera (lidocaine 70mg/tetracaine 70mg): All subjects received 2 patch applications, one Synera and one placebo. These 2 patch applications were done on separate days. Subjects in this arm received Synera patch for the first application (day 1), and then placebo for the second (day 2 or after).
- Placebo First, Then Synera: Synera (lidocaine 70mg/tetracaine 70mg): All subjects received 2 patch applications, one Synera and one placebo. These 2 patch applications were done on separate days. Subjects in this arm received placebo patch for the first application (day 1), and then Synera for the second (day 2 or after).
Period: Overall Study
Arm/Group | Synera First, Then Placebo | Placebo First, Then Synera
Started | 32 | 29
Completed | 28 | 26
Not Completed | 4 | 3
Not completed — Received 1 patch | 2 | 1
Not completed — No patch received | 2 | 2

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Synera First, Then Placebo | Placebo First, Then Synera | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.2) | 60.3 (13.0) | 60.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 12 | 15 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31 | 24 | 55
  African American | 1 | 4 | 5
  Indian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With No or Minor Pain (VAS<3)
Description: The primary efficacy endpoint is the subject's report of pain intensity regarding the venipuncture using a 0-10 VAS. The VAS <3 is considered as patients with no or minor pain and would be compared between 2 groups.
Time Frame: 30 minutes after the venipuncture.
Population: Normal completion patients.
Measure: Number; unit: percentage of participants
Groups:
- Synera: Treated with Synera.
- Placebo: Treated with Placebo.
Arm/Group | Synera | Placebo
Number analyzed (Participants) | 54 | 54
percentage of participants | 38.0 | 21.3

2. Primary Outcome: Percentage of Patients With No Pain (VAS=0)
Description: The primary efficacy endpoint is the subject's report of pain intensity regarding the venipuncture using a 0-10 VAS. The VAS =0 is considered as patients with no pain and would also be compared between 2 groups.
Time Frame: 30 minutes after the venipuncture.
Population: Normal completion patients
Measure: Number; unit: percentage of participants
Arm/Group | Synera | Placebo
Number analyzed (Participants) | 54 | 54
percentage of participants | 19.4 | 8.3

3. Secondary Outcome: Global Assessment of Satisfaction With Venipuncture
Description: Rates of Satisfied and very satisfied are used to be compared between two groups.
Time Frame: 30 minutes after the venipuncture.
Population: Normal completion patients
Measure: Number; unit: percentage of participants
Arm/Group | Synera | Placebo
Number analyzed (Participants) | 54 | 54
percentage of participants | 74.0 | 53.7

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Synera | Placebo
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 25/54 | 18/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synera (N=54) | Placebo (N=54)
VERY SLIGHT ERYTHEMA (Skin and subcutaneous tissue disorders) | 11 (11) | 11 (11)
WELL-DEFINED ERYTHEMA (Skin and subcutaneous tissue disorders) | 14 (14) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No